CLINICAL TRIAL: NCT04080050
Title: A Long-term Follow-up Study to Evaluate the Safety and Efficacy of RGX-501
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RGX-501-102
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Homozygous Familial Hypercholesterolemia (HoFH)
Keywords: LDL Receptors; Gene Therapy; Metabolic Diseases; Rare Diseases; Genetic Diseases; Atherosclerosis; Cardiovascular Disease
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia; Hyperlipoproteinemia Type II; Metabolic Diseases; Rare Diseases; Genetic Diseases, Inborn; Atherosclerosis; Cardiovascular Diseases | interventions — Genetic Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RGX-501: Study participants who have received RGX-501 gene therapy in a separate parent trial
  Interventions: Drug: Single intravenous (IV) dose of human Low Density Lipoprotein Receptor (LDLR) Gene Therapy

INTERVENTIONS:
Drug: Single intravenous (IV) dose of human Low Density Lipoprotein Receptor (LDLR) Gene Therapy — No investigational product will be administered in this study. All participants have previously received a one-time intravenous infusion of RGX-501 in a separate clinical trial
  Other Names: RGX-501

SUMMARY:
This long-term observational study is designed to follow subjects who, during another Clinical Study, received gene therapy treatment used to treat their Homozygous Familial Hypercholesterolemia (HoFH) disease. This study is intended to follow those subjects for up to 5 years since they received treatment to look for any long-term safety concerns. There is no investigational drug or therapy provided as part of this study.

DETAILED DESCRIPTION:
Homozygous Familial Hypercholesterolemia (HoFH) is a rare genetic metabolic disorder characterized by absent or severely reduced capacity to catabolize circulating LDL particles by the hepatic LDL receptor. As a consequence, HoFH subjects present abnormal total plasma cholesterol (LDL-C) levels, resulting in severe atherosclerosis often leading to early onset of cardiovascular disease. Early initiation of aggressive treatment for these patients is therefore essential. Unfortunately, despite existing therapies, treated LDL-C levels could remain well above acceptable levels. Thus, the functional replacement of the defective LDLR via AAV-based liver-directed gene therapy, RGX-501, may be a viable approach to treat this disease and improve response to current lipid-lowering treatments.

This is a prospective, observational study to evaluate the long-term safety and efficacy after a single administration of RGX-501. Eligible participants are those who previously have enrolled in a clinical study and received a single intravenous infusion of RGX-501.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this study, a participant must have previously received RGX-501 in a separate parent trial, and the participant or participant's legal guardian(s) is/(are) willing and able to provide written, signed informed consent after the nature of the study has been explained, prior to any research-related procedures.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have previously received RGX-501 in a separate parent trial
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2024-09-29 (Estimated); Study Completion 2025-09-29 (Estimated)

PRIMARY OUTCOMES:
Number of incidents of new and unexpected adverse events and serious adverse events. | Up to 5 years after receiving treatment with RGX-501
  The number of times a new and unexpected adverse event and/or serious adverse event is reported.

SECONDARY OUTCOMES:
The absolute LDL-C level in mg/dL by beta quantification | Year 3 after receiving treatment with RGX-501
  Absolute LDL-C level by beta quantification at Year 3 after receiving treatment with RGX-501
Absolute total cholesterol, LDL-C, very low density lipoprotein cholesterol (VLDL-C), high density lipoprotein cholesterol (HDL-C), calculated non-HDL-C, triglycerides (TG), and lipoprotein a (Lp(a)) over the study duration | Up to 5 years after receiving treatment with RGX-501
  Absolute total cholesterol, LDL-C, very low density lipoprotein cholesterol (VLDL-C), high density lipoprotein cholesterol (HDL-C), calculated non-HDL-C, triglycerides (TG), and lipoprotein a (Lp(a)) over the study duration
Usage of lipid-lowering therapies over time | Up to 5 years after receiving treatment with RGX-501
  Usage of lipid-lowering therapies over time

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - Columbus Location, Columbus, Ohio
  - Portland location, Portland, Oregon
  - Philadelphia location, Philadelphia, Pennsylvania
  - Nashville location, Nashville, Tennessee
- Montreal location, Montreal, Quebec, Canada
- Rotterdam location, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No